CLINICAL TRIAL: NCT02604186
Title: Botulinum Toxin in Patients With Hereditary Spastic Paraplegia: a Randomized, Double-blind, Placebo-controlled, Crossover Study
Brief Title: Effects of Botulinum Toxin Injections in Patients With Hereditary Spastic Paraplegia
Acronym: SPASTOX
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Cristália Produtos Químicos Farmacêuticos Ltda. (Industry)
Responsible Party: Principal Investigator, Marcondes Cavalcante França Júnior, MD, Phd, University of Campinas, Brazil
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAAE: 48177315.9.1001.5404
Record Dates: First submitted 2015-11-09; First posted 2015-11-13 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Hereditary Spastic Paraplegia
Keywords: Spasticity; Botulinum Toxin; Hereditary Spastic Paraplegia
MeSH Terms: conditions — Spastic Paraplegia, Hereditary; Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum Toxin Injections (Experimental): Botulinum Toxin injections at adductors and triceps surae
  Interventions: Other: Botulinum Toxin Injections
- Placebo Injections (Placebo Comparator): Placebo injections at adductors and triceps surae
  Interventions: Other: Placebo Injections

INTERVENTIONS:
Other: Botulinum Toxin Injections — Each patient in the treatment group will receive 400 units of botulinum toxin. 100 units will be injected at adductors at each leg and 100 units will be applied in each triceps surae bilaterally.
  Arms: Botulinum Toxin Injections
Other: Placebo Injections — Each patient in the placebo group will receive sterile sodium chloride injections at adductors and triceps surae muscles bilaterally.
  Arms: Placebo Injections

SUMMARY:
Hereditary spastic paraplegias constitute a heterogeneous group of diseases with the common predominant feature of spasticity of the lower limbs. The clinical picture is composed of difficulty walking, exaggerated deep reflexes, pathological reflexes such as the Babinski sign, sphincter disturbances and various degrees of weakness as well as sensory disturbances.

Spasticity is the symptom that provoques greater incapacity. Although there have been recent advances in the genetic and pathogenic characterization of SPG there is scarcity of therapeutic options. The Botulinum Toxin (BTx) is a well established treatment for movement disorders such as cervical dystonia, blepharospasm, and arm spastic following stroke.

Therefore, the investigators propose the execution of a randomized, double-blind, placebo-controlled, crossover study to evaluate the efficacy of the treatment with Btx over SPG patient's gait. The primary outcome measure will be gait velocity with the 10 meter walking test 8 weeks after injection. Each participant will be submitted to one injection session of Btx and one of placebo (consisting of sterile sodium chloride), each one separated by a period of 6 months. The primary and secondary outcomes will be evaluated by a blind investigator 8 weeks after each injection session.

DETAILED DESCRIPTION:
Introduction

Hereditary spastic paraplegias (SPG) constitute a heterogeneous group of diseases with a common predominant feature: spasticity of the lower limbs and difficulty walking. The neurologic examination reveals spasticity, exaggerated and pathological reflexes, such as the Babinski sign, and minor hypoesthesia. Spasticity is more evident when the patient walks than during passive movement. Weakness may or may not be present, and typically is less disabling than spasticity, especially during the initial years of the disease. The increase in tonus leads to reduced amplitude of movement and abnormal posture, altogether leading to a very slow gait, falls and articular deformities. Clinically, SPG is divided into pure and complicated forms. The first one is characterized by almost exclusive dysfunction of the pyramidal tracts. Minor sensory and sphincter disturbances are also present. The complicated subtypes encompass a wide variety of associated features such as ataxia, cognitive decline and vision loss. Genetically, SPGs are divided into autosomal dominant, autosomal recessive and X-linked forms. Pure forms are mostly inherited in an autosomal dominant manner, whereas the autosomal recessive forms mostly manifest as complicated forms. Although useful clinically, this genotype-phenotype correlation is not always true. The most used SPG classification is based on the locus that harbors the mutated gene. Each subtype is designated by the initials SPG, followed by a number that corresponds to a specific gene. The gene number is established following the chronological order of identification of each locus.

The discovery of new genes and the unraveling of molecular pathways of SPGs have lead to a better understanding of the disease in the past few years. Despite that, there are very few treatment options . There is no placebo-controlled clinical trial performed to assess any therapeutic intervention for SPG. Oral anti-spastic agents such as baclofen and tizanidine are frequently employed. When the response is inadequate, or there are significant side effects, botulinum toxin injections may be attempted. The substance blocks liberation of acetylcholine from the pre-synaptic cleft. With less activation of the nicotinic receptors at the post-synaptic junction the muscle contraction is inhibited. Botulinum Toxin (Btx) is a first-line treatment for movement disorders such as cervical dystonia, blepharospasm, and spastic arm following stroke. Studies with Btx in patients with SPG are limited to small open-label case series, and there is no solid evidence that patients actually benefit from this therapy. The rationale basis for its use is based on the well established knowledge that Btx reduces muscle tonus. The functional impact on gait, on the other hand, is not well known, as well as the impact this treatment could produce over symptoms such as fatigue and pain.

Justification Spasticity is the most disabling manifestation in patients with SPG. Although there have been recent advances in the genetic and pathogenic characterization of the disease, there is scarcity of therapeutic options. The use of oral anti-spastics is limited by frequent side effects such as somnolence and drowsiness. Therefore, the investigators designed a randomized, double-blind, placebo-controlled, crossover trial to evaluate the efficacy and safety of Btx injections in patients with SPG. The primary outcome measure will be gait velocity assessed through the 10 meter walking test 8 weeks after injection. Each participant will be submitted to one injection session with Btx and one with placebo (consisting of sterile sodium chloride), each one separated by a period of 6 months.

Objectives General Objective To evaluate the effects of Btx compared to placebo injections in a cohort of patients with SPG. The primary outcome will be increase in gait velocity, a measure that reflects functional gain. Secondary outcomes will include measures of spasticity, pain and fatigue.

Specific Objectives

* To investigate whether Btx injections improve maximum gait velocity in patients with SPG compared to injections of placebo.
* To investigate the effects of the treatment versus placebo over the following functional measures: Spastic Paraplegia Rating Scale (SPRS), Visual Analogic Pain Scale, Brief Pain inventory, Modified fatigue impact scale, Ashworth Spasticity and muscle strength (through the Medical Research Council Scale) for adductors and triceps surae muscles.

Methods Patients Selection Patients will be selected during regular consultations at two University Hospitals in Brazil: the University of Campinas (UNICAMP) and the Federal University of Paraná (UFPR).

Sample size Estimate The sample size calculus was based on a recent exploratory study (Niet, 2015) where 15 patients with autosomal dominant spastic paraplegia were submitted to Btx injections at the triceps surae. This provoked and increase in gait velocity of 9% after 4 weeks and of 12% after 18 weeks. Estimating a 12% effect for an alfa value of 0.08 and a p value of 0.05, the investigators obtained a N of 54 individuals after correcting for possible losses (approximately 10%). The Stata version 13.1 was used for the estimates.

Procedures All patients recruited will be randomized to receive injections of Prosigne (Botulinum Toxin A) or a Placebo solution (sterile Sodium Chloride 0.9%). Each patient in the treatment group will receive 400 units of botulinum toxin. 100 units will be injected at adductors at each leg and 100 units will be applied in each triceps surae bilaterally. The botulinum toxin as well as the placebo solutions will be prepared by a blind investigator. Prosigne will be diluted with sterile sodium chloride (10U/0.2mL). Within 24 to 28 weeks of the first treatment groups will be switched. Those patients that received botulinum toxin will receive a placebo solution and vice-versa (crossover point). During the study, all patients will be oriented to maintain the ongoing use of medications. They will receive an explanatory sheet regarding stretching exercises, at least one month before receiving treatment, and will be trained by a physiotherapist to execute those exercises twice a week.

Data analysis and interpretation Patients will be evaluated by an experienced and blind neurologist regarding the efficacy parameters of the study. This evaluation will take place immediately before each treatment section and 8 weeks after it. The primary outcome measure will be maximum gait velocity. Each patient will be asked to walk a 10 meter distance barefooted 3 times, as fast as he can. The average velocity between the 3 trials will be used as the final measure. Assistive devices are permitted. Spastic Paraplegia Rating Scale (SPRS), Ashworth modified spasticity scale, medical research council scale for muscular strength (for adductors, thigh and triceps surae muscle groups), visual analogic scale of pain, brief pain inventory and the modified fatigue impact scale, together with the 10 meter comfortable walking velocity, will be evaluated at the same day as the primary outcome measure and will serve as secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* Clinical diagnosis of Hereditary Spastic Paraplegia
* Ability to walk at least 10 meters: Assistive devices are permitted

Exclusion Criteria:

* Wheelchair bound patients
* Additional neurological symptoms that may significantly impact gait such as ataxia, polyneuropathy or dementia.
* Fixed tendon contractures
* Antecedents of allergy or adverse reaction to botulinum toxin
* Pregnancy or breastfeeding condition
* Mental retardation
* Dementia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-03-09 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in 10 meter maximum gate velocity | 8 weeks after injections
  The primary outcome measure will be change from baseline in maximum gait velocity. Each patient will be asked to walk a 10 meter distance barefooted 3 times, as fast as he can. The average velocity between the 3 trials will be used as the final measure. Assistive devices are permitted.

SECONDARY OUTCOMES:
Change from baseline in Spastic Paraplegia Rating Scale (SPRS), | 8 weeks after each procedure
  The same neurologist will examine the patient to evaluate change at the SPRS scale
Change from baseline in Ashworth spasticity scale of adductors and triceps surae muscles | 8 weeks after each procedure
  The same neurologist will examine the patient to evaluate change from baseline
Change from baseline in muscle strengh (Medical Research Council scale) concerning adductors and triceps surae muscles. | 8 weeks after each procedure
  The same neurologist will examine the patient to evaluate change from baseline
Change from baseline in visual analogic scale of pain | 8 weeks after each procedure
  this scale will be applied by a neurologic physiotherapist
Change from baseline in brief pain inventory scale | 8 weeks after each procedure
  this scale will be applied by a neurologic physiotherapist
Change from baseline in modified fatigue impact scale | 8 weeks after each procedure
  this scale will be applied by a neurologic physiotherapist
Change from baseline in 10 meter comfortable walking velocity | 8 weeks after each procedure
  this scale will be applied by a neurologic physiotherapist

CONTACTS AND LOCATIONS:
Overall Officials: Marcondes c França Júnior, M.D, PhD, Principal Investigator — University of Campinas, Brazil
Locations (1):
- Univeristy of Campinas Hospital, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Niet M, de Bot ST, van de Warrenburg BP, Weerdesteyn V, Geurts AC. Functional effects of botulinum toxin type-A treatment and subsequent stretching of spastic calf muscles: a study in patients with hereditary spastic paraplegia. J Rehabil Med. 2015 Feb;47(2):147-53. doi: 10.2340/16501977-1909. PMID 25325386